CLINICAL TRIAL: NCT06147609
Title: Effect of Fixed and Removable Space Maintainer on Some Salivary Parameters: An In-Vivo Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: space maintainers and saliva
Record Dates: First submitted 2023-11-17; First posted 2023-11-27 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Premature Loss of Primary Teeth
Keywords: Teeth loss; Missing teeth
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- children with lower lingual holding arch space maintainer (Active Comparator): non functional fixed space maintainer used in the mandibular arch to maintain arch length by prevention of mesial movement of permanent first molar
  Interventions: Device: lower lingual holding arch space maintainer
- children with removable partial denture space maintainer (Active Comparator): functional Removable space maintainer that not only maintain the mesiodistal space, but vertical dimension and masticatory function is also assured
  Interventions: Device: Removable partial denture space maintainer

INTERVENTIONS:
Device: lower lingual holding arch space maintainer — lower lingual holding arch space maintainer is an orthodontic device which connects two molars lower dental arch. it has an archwire, adapted to the lingual side of the lower anterior teeth, that soldered to the bands on first permanent molar
  Arms: children with lower lingual holding arch space maintainer
Device: Removable partial denture space maintainer — Removable Partial Denture consists of a pink or gum-colored plastic base to which the new, artificial, replacement teeth are attached to. a metal framework holds the denture in place inside the mouth
  Arms: children with removable partial denture space maintainer

SUMMARY:
The aim of this study is to evaluate and compare the effect of lower lingual holding arch space maintainer versus removable partial denture space maintainer on some salivary parameters (salivary flow rate, pH, viscosity and buffering capacity).

DETAILED DESCRIPTION:
This study is a randomized clinical trial, it will be conducted on forty children, aged from (7-10) years, who are in need for space maintainer.

* Children will be randomly and equally divided into two groups according to type of space maintainer used; group (1): twenty children with lower lingual holding arch, group (2): twenty children with removable partial denture.
* Un-stimulated and stimulated saliva will be collected at specific duration of time from children before the delivery of the appliance and after 1, 3 and 6 months of wearing the space maintainer to measure salivary flow rate, pH, viscosity and buffering capacity.

ELIGIBILITY:
Inclusion Criteria:

Apparently healthy with no systemic disease. Age between 7-10 years old. Both boys and girls will be included.

Children with the following dental criteria:

Clinical criteria:

* Children should have a good oral hygiene.
* Children in mixed dentition stage.
* Fully erupted permanent lower first molar.
* Children with multiple loss of deciduous molar teeth.
* Seek for space maintainer appliance.

Radiographic criteria :

* Presence of at least 1mm bone overlaying successor.
* Tooth germ with less than one third of the root formed.

Exclusion Criteria:

* Allergy to any used material

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of salivary flow of un-stimulated saliva | before delivery of appliance, after 1 month, 3 months, 6 months
  Un-stimulated whole saliva will be collected from all individuals by direct expectoration into a sterile container over a period of 10 min by spitting method, so that the flow rate could be calculated by dividing the amount of expectorated saliva by 10 min
Assessment of salivary flow of stimulated saliva | before delivery of appliance, after 1 month, 3 months, 6 months
  To stimulate saliva, the subjects will be asked to chew a piece of paraffin wax, and saliva will be collected for 5 min in a measuring cup with 1ml gradation marks; the stimulated salivary flow rate (ml/min) will be calculated by dividing the amount of expectorated saliva by 5 min
Assessment of Salivary pH | before delivery of appliance, after 1 month, 3 months, 6 months
  Salivary pH will be measured using an electronic pH meter
Assessment of viscosity of saliva | before delivery of appliance, after 1 month, 3 months, 6 months
  Salivary viscosity will be determined by allowing saliva to flow through a tube of circular cross section to measure the flow rate . This will be done using the Ostwald viscometer.
Assessment of buffering capacity | before delivery of appliance, after 1 month, 3 months, 6 months
  By estimating the pH change after HCl titration into un-stimulated saliva for a buffering capacity test.

CONTACTS AND LOCATIONS:
Overall Officials: Yousra S Mohamed, PhD, Principal Investigator — Lecturer
Locations (1):
- Faculty of medicine, Suez Canal University, Ismailia, Egypt

REFERENCES:
- [Background] Alessandri Bonetti G, Incerti Parenti S, Garulli G, Gatto MR, Checchi L. Effect of fixed orthodontic appliances on salivary properties. Prog Orthod. 2013 Jun 18;14:13. doi: 10.1186/2196-1042-14-13. PMID 24326149
- [Background] Charan J, Biswas T. How to calculate sample size for different study designs in medical research? Indian J Psychol Med. 2013 Apr;35(2):121-6. doi: 10.4103/0253-7176.116232. PMID 24049221
- [Background] Dallel I, Ben Salem I, Merghni A, Bellalah W, Neffati F, Tobji S, Mastouri M, Ben Amor A. Influence of orthodontic appliance type on salivary parameters during treatment. Angle Orthod. 2020 Jul 1;90(4):532-538. doi: 10.2319/082919-562.1. PMID 33378497
- [Background] Essawy K., Gomaa Y. & Khattab N. (2021). 'Clinical Performance of CAD /CAM Fixed Functional Space Maintainer Made of Poly Ether Ether Ketone (PEEK)'. Minia Journal of Medical Research, 32(4): pp.7-12. doi: 10.21608/mjmr.2021.241647
- [Background] Govindaraj S., Daniel M., & Vasudevan S. & Kumaran J. (2019). 'Changes in Salivary Flow Rate, pH, and Viscosity Among Working Men and Women'. Dentistry and Medical Research, 7(2): pp. 56-59. doi:10.4103/dmr.dmr_20_19.
- [Background] Kandhan T., Jeevanandan G. & Rajasekar A. (2019). 'Prevalence of Lingual Arch Space Maintainer Among Children Between the Age Groups Of 6-10 Years - A Retrospective Study'. International Journal of Dentistry and Oral Science, 8(5): pp. 21-25. doi:10.19070/2377-8075-SI02-08005.
- [Background] Kizilci E., Arikan V., Ozalp N. & Ozcelik B. (2021) 'The Effect of Space Maintainers on Salivary pH, Flow Rate, and the Oral Microflora'. Australasian Orthodontic Journal, 37(2): pp.259-264. doi:10.21307/aoj-2021.028
- [Background] Kukreja P, Hugar SM, Hallikerimath S, Sogi S, Badakar C, Thakkar P. Evaluation of the Effect of Fixed and Removable Appliances on Salivary Parameters (Salivary Flow Rate pH and Buffering Capacity) in Children Aged 5-12 Years: An In Vivo Study. Int J Clin Pediatr Dent. 2021 Nov-Dec;14(6):774-778. doi: 10.5005/jp-journals-10005-2066. PMID 35110870
- [Background] Moritsuka M, Kitasako Y, Burrow MF, Ikeda M, Tagami J. The pH change after HCl titration into resting and stimulated saliva for a buffering capacity test. Aust Dent J. 2006 Jun;51(2):170-4. doi: 10.1111/j.1834-7819.2006.tb00422.x. PMID 16848266
- [Background] Mosharrafian S, Baghalian A, Hamrah MH, Kargar M. Clinical Evaluation for Space Maintainer after Unilateral Loss of Primary First Molar in the Early Mixed Dentition Stage. Int J Dent. 2021 Dec 27;2021:3967164. doi: 10.1155/2021/3967164. eCollection 2021. PMID 34987584
- [Background] Ramakrishnan M, Dhanalakshmi R, Subramanian EMG. Survival rate of different fixed posterior space maintainers used in Paediatric Dentistry - A systematic review. Saudi Dent J. 2019 Apr;31(2):165-172. doi: 10.1016/j.sdentj.2019.02.037. Epub 2019 Feb 14. PMID 30983825
- [Background] Sathyaprasad S, Krishnareddy MG, Vinod V, Das N, Ramesh R, Ilyas I. Comparative Evaluation of Fixed Functional Cantilever Space Maintainer and Fixed Nonfunctional Space Maintainer: A Randomized Controlled Trial. Int J Clin Pediatr Dent. 2022 Nov-Dec;15(6):750-760. doi: 10.5005/jp-journals-10005-2478. PMID 36866140
- [Background] Sethuraman G., Daniel M., Vasudevan S. & Kumaran J. (2019). 'Changes in Salivary Flow Rate, pH, and Viscosity among Working Men and Women'. Dentistry and Medical Research, 7(2): pp. 56-59. doi: 10.4103/dmr.dmr_20_19
- [Background] Srivastava V.(2011). 'Modern Pediatric Dentistry '.1 st edition. Jaypee Brothers Medical Publishers (P) Ltd, India: pp. 95-99